CLINICAL TRIAL: NCT07143344
Title: The Effect of Fermented Lingonberry Spray on Oral Health - The Pilot Study
Brief Title: This Study Utilized Fermented Lingonberry Juice in a Spray Form, Allowing it to be Applied to the Mouth Four Times a Day.
Acronym: FLJS_TRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahanna oy (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LING_TRE; TYH2022225 (Other Grant/Funding Number: University of Helsinki); TYH 2024332 (Other Grant/Funding Number: University of Helsinki); TYH 2025382 (Other Grant/Funding Number: University of Helsinki); Y2519SU010 (Other Grant/Funding Number: University of Helsinki)
Record Dates: First submitted 2025-08-12; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Bleeding on Probing; Pocket Depth; Plaque Control; Saliva Microbiome
Keywords: fermented lingonberry juice; saliva test; mouthrinse; aMMP-8 test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients were randomly selected from a private dental clinic in Tampere, Finland for the study (Experimental): Participants used approximately ten sprays four times a day (approx. 5,5 ml/ day) of FLJ-spray (Lingora® Oral Spray, Berries United Ltd, Helsinki, Finland) for a month.
  Interventions: Other: Fermented lingonberry juice sprey

INTERVENTIONS:
Other: Fermented lingonberry juice sprey — Patented fermented lingonberry juice sprey
  Other Names: FLJ; fermented lingonberry juice

SUMMARY:
A human intervention study was performed to examine the antimicrobial effects of fermented lingonberry spray (FLJ spray) treatment, used for a period of 30 days.

DETAILED DESCRIPTION:
Traditional clinical oral examinations, periodontal status and sample gatherings were performed at start point, two and four weeks. Bleeding on probing (BOP), visible plaque index (VPI), probing pocket depths (PPD) were examined and active-matrix metalloproteinase - 8 (aMMP-8) mouthrinse assays (Cutt-off 20 ng/ml) were carried out. Additionally, stimulated and resting saliva, pH and buffering capacity were tested as saliva test. A questionnaire assessing dry mouth symptoms was also recorded from the patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients or patients with systemic diseases with good cognitive abilities
* with or without xerostomia.

Exclusion Criteria:

* use of other mouthwash products, including chlorhexidine
* current use of antibiotics.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
The effects of fermented lingonberry spray in the mouth. | Up to one month
  Changes of bleeding on probing (BOP), from six measurement point, visible plaque index (VPI), score 1-3, probing pocket depths (PPD) and active-matrix metalloproteinase - 8 (aMMP-8) mouthrinse assays (Cutt-off 20 ng/ml), numerical value were carried out to one month.
the time points on the levels of each salivary parameter were determined with the repeated measures ANOVA analysis. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Helsinki, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial.
Supporting Information: Study Protocol, CSR